CLINICAL TRIAL: NCT07349017
Title: A Single-Center, Randomized, Blinded Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of Influenza Virus Vaccine (BK-01 Adjuvant) in Populations Aged 18 Years and Older
Brief Title: A Phase I Trial to Evaluate the Safety and Immunogenicity of Influenza Virus Split Vaccine (Adjuvant)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun BCHT Biotechnology Co. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: B1701-F20240612-1
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- influenza vaccine（BK01 adjuvant） (Experimental)
  Interventions: Biological: influenza vaccine（BK01 adjuvnat）
- approved influenza vaccine (Active Comparator)
  Interventions: Biological: approved influenza vaccine
- adjuvant placebo (Placebo Comparator)
  Interventions: Biological: adjuvant placebo
- placebo (Placebo Comparator)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: influenza vaccine（BK01 adjuvnat） — Each human dose is 0.5 mL, containing 15 μg of hemagglutinin from each type of influenza virus strain.
  Arms: influenza vaccine（BK01 adjuvant）
Biological: approved influenza vaccine — Each human dose is 0.5 mL, containing 15 μg of hemagglutinin from each type of influenza virus strain.
  Arms: approved influenza vaccine
Biological: adjuvant placebo — Each human dose is 0.5 mL, containing no influenza virus strain hemagglutinin. The main ingredient is BK-01 adjuvant.
  Arms: adjuvant placebo
Biological: placebo — Each human dose is 0.5 mL. The main ingredient is sodium chloride.
  Arms: placebo

SUMMARY:
The goal of this clinical trial is to evaluate the safety and immunogenicity of the influenza virus vaccine (BK-01 adjuvant) in people aged 18 years and older.

The main questions it aims to answer is:

• Incidence rate of adverse reactions/events after administration Participants will be randomly vaccinated with a single dose of the trial vaccine, control vaccine, adjuvant placebo, or placebo in a 1:1:1:1 ratio. After vaccination, all participants will undergo up to 30-day observation and blood collection.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years and above;
* Have not received any influenza vaccine in the past six months and have no plan to receive other influenza vaccines during the trial period;
* Have not had influenza in the past 6 months (confirmed by any clinical, serological, or microbiological method);
* Able to obtain the participant's own informed consent;
* The participant themselves can comply with the requirements of the clinical trial protocol.

Exclusion Criteria:

* Axillary temperature > 37.0℃ on the day of enrollment;
* Female participants of childbearing age with a positive urine pregnancy test result, or who are breastfeeding, or have a plan to have children within 12 months;
* Those with a history of severe allergic diseases (such as anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergic necrotic reaction), or who are allergic to any component of the test vaccine, such as eggs, gentamicin sulfate, formaldehyde, TritonX-100, etc.;
* Those with clinically significant abnormal laboratory test results, which are determined by the researcher as unsuitable for vaccine vaccination；
* Those who have had an acute illness, acute exacerbation of a chronic disease, or used antipyretic, analgesic, or anti-allergic drugs within the past 3 days;
* Autoimmune diseases or immune deficiency, asplenia, functional asplenia, and asplenia or splenectomy caused by any condition; those who have received long-term systemic drugs within the past 3 months or plan to receive long-term systemic drugs during the trial, including immunosuppressive and/or immunomodulatory drugs, leukotoxic therapy, etc. (for more than 14 consecutive days);
* Those with congenital malformations affecting organ function, Down's syndrome, major diseases or major potential diseases that may interfere with or hinder the completion of the trial (such as: severe cardiovascular or chronic diseases in the decompensated stage, cor pulmonale, pulmonary edema, severe liver and kidney diseases, severe or symptomatic diabetes, current malignant tumors, etc.);
* Those with uncontrolled hypertension with drugs (18-59 years old: systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg; ≥ 60 years old: systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg);
* Those with a history or family history of mental and neurological diseases such as convulsions, epilepsy, encephalopathy, and psychosis; Those with contraindications to intramuscular injection and blood collection, such as: diagnosed with sickle cell anemia, thrombocytopenia, any coagulation disorder, or receiving anticoagulant therapy, etc.;
* Those who have received blood products or immunoglobulin products within 3 months before receiving the test vaccine or plan to use them during the trial;
* Those who have received other clinical trial drugs within 1 month before receiving the test vaccine or are participating in other clinical trials, received live attenuated vaccines, viral vector vaccines, or nucleic acid vaccines within 14 days, or received subunit, recombinant, or inactivated vaccines within 7 days;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-02-07 (Estimated); Primary Completion 2026-04-25 (Estimated); Study Completion 2027-03-07 (Estimated)

PRIMARY OUTCOMES:
Safety outcome | upto 30 days after vaccination
  Incidence rate of adverse reactions/events

SECONDARY OUTCOMES:
Immunogenicity outcome | upto 30 days after vaccination
  seroconversion rate of HI antibody
Immunogenicity outcome | upto 30 days after vaccination
  HI antibody titers

IPD SHARING:
Plan to Share IPD: Yes